CLINICAL TRIAL: NCT03913351
Title: Lifestyle Modification Programme for HIV-infected Individuals With Non-alcoholic Fatty Liver Disease: A Randomized Controlled Trial
Brief Title: Lifestyle Modification Programme for HIV-infected Individuals With Fatty Liver
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Study Protocol LSM V2
Record Dates: First submitted 2019-04-09; First posted 2019-04-12 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: NAFLD; Hiv
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle modification program (Experimental): The dietary intervention program will be scheduled for 12 months, and conducted by a dietitian.The program aims to increase energy expenditure and reduce caloric intake, with an emphasis on long-term lifestyle and behavioural change. An exercise instructor will provide advice on physical activity. A mobile tracking device to monitor calories expenditure will be provided to each participant during they study period to encourage physical activity.
  Interventions: Behavioral: Lifestyle modification
- Control (No Intervention): standard care of treatment, as in routine clinical practice

INTERVENTIONS:
Behavioral: Lifestyle modification — The program consists of education on glycemic index, balanced diet, interpretation of food labels, food exchanges, healthy eating out techniques and healthy cooking methods.
  Arms: Lifestyle modification program

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) is rising in prevalence, and will likely become the predominant cause of chronic liver disease in HIV-infected individuals.

Metabolic factors and obesity are important risk factors for NAFLD in HIV-infected individuals. There is currently no approved effective pharmacological treatment for fatty liver disease. Therefore, lifestyle modification directing at weight loss is currently the cornerstone of treatment for fatty liver disease in the general population. Hypocaloric diets can improve fatty liver in the general population, but the most effective specific dietary interventions are yet to be elucidated.

The study aims to 1. determine the efficacy of a lifestyle modification programme in inducing resolution of NAFLD in HIV-infected individuals 2. to determine the efficacy of a lifestyle modification programme in improving insulin resistance, pro-inflammatory markers, and liver fibrosis in HIV-infected individuals with fatty liver disease 3. to determine changes in intestinal microbiome secondary to the lifestyle modification programme, and the association with resolution of NAFLD in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or above
* positive HIV antibody, on anti-retroviral therapy
* HIV viral load ≤50 copies/mL for ≥6 months
* intrahepatic triglyceride content ≥5% on magnetic resonance spectroscopy

Exclusion Criteria:

* current AIDS-defining illness
* active malignancy, or history of malignancy within the last 5 years
* hepatitis B and/or hepatitis C co-infection, as determined by positive HBsAg and anti--HCV antibody
* alcohol consumption >30g per week in men or 20g per week in women
* alanine aminotransferase (ALT) above 10 times the upper limit of normal
* liver decompensation (as evidenced by bilirubin above 50 µmol/l, platelet count below 100 × 109/l, prothrombin time above 1.3 times the upper limit of normal, albumin below 35 g/l, presence of ascites or varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Resolution of NAFLD | 12 months
  The primary endpoint is the proportion of patients with resolution of NAFLD as determined by proton-magnetic resonance spectroscopy at month 12.

SECONDARY OUTCOMES:
Partial resolution of NAFLD | 12 months
  Partial resolution of NAFLD is defined as absolute reduction of hepatic triglyceride content by 30% or more.
Changes in adiposity | 12 months
  The changes in visceral fat will be determined by magnetic resonance imaging at the same session
Change in liver fibrosis | 12 months
  The changes in liver fibrosis will be determined by transient elastography by Fibroscan
Metabolic endpoints | 12 months
  The proportion of patients with impaired fasting glucose will be determined
Metabolic endpoints | 12 months
  The proportion of patients with diabetes will be determined
Metabolic endpoints | 12 months
  The proportion of patients with insulin resistance (estimated by the homeostasis model) will be determined
Metabolic endpoints | 12 months
  The proportion of patients with hypertension will be determined
Metabolic endpoints | 12 months
  The proportion of patients with dyslipidemia will be determined
Metabolic endpoints | 12 months
  The proportion of patients with metabolic syndrome will be determined
Biomarkers of inflammation and monocyte activation | 12 months
  Changes from baseline in adipokines (adiponectin and leptin)
Biomarkers of inflammation and monocyte activation | 12 months
  Changes from baseline in marker of endothelial cell activation (ICAM-1)
Biomarkers of inflammation and monocyte activation | 12 months
  Changes from baseline in marker of monocyte activation (sCD163)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Derived] Li G, Wong VW, Chan RS, Sin DM, Chu W, Wong V, Cheung C, Lam S, Lin H, Yeung S, Li TC, Ho TH, Wong GL, Yip TC, Lui GC. Lifestyle modification programme for people living with HIV with metabolic dysfunction-associated steatotic liver disease: a randomised controlled trial. Lancet HIV. 2025 Jun;12(6):e416-e427. doi: 10.1016/S2352-3018(25)00032-3. Epub 2025 May 8. PMID 40347962